CLINICAL TRIAL: NCT03581123
Title: Spinal Manipulation and Patient Self-Management for Preventing Acute to Chronic Back
Brief Title: Spinal Manipulation and Patient Self-Management for Preventing Acute to Chronic Back Pain
Acronym: PACBACK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: University of Pittsburgh (Other); University of Washington (Other); University of North Texas Health Science Center (Other); Oregon Health and Science University (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CSH-2018-26524
Record Dates: First submitted 2018-05-03; First posted 2018-07-10 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Acute Pain; Low Back Pain, Mechanical
Keywords: acute/subacute low back pain; randomized clinical trial; self-management; behavioral modification; spinal manipulation therapy; standard medical care; secondary prevention
MeSH Terms: conditions — Acute Pain; Low Back Pain | interventions — specific substance maruyama

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Supported-Self management (SSM) (Experimental): Supported-Self management
  Interventions: Behavioral: Supported-Self Management (SSM)
- Spinal Manipulation Therapy (SMT) (Experimental): Spinal Manipulation Therapy
  Interventions: Other: Spinal Manipulation Therapy (SMT)
- SMT + SSM (Experimental): Spinal Manipulation Therapy + Supported Self-Management
  Interventions: Combination Product: SMT + SSM
- Standard Medical Care (SMC) (Active Comparator): Standard Medical Care
  Interventions: Drug: Standard Medical Care (SMC)

INTERVENTIONS:
Behavioral: Supported-Self Management (SSM) — Provides low back pain sufferers opportunities to develop the capacity and motivation to self-manage their pain in an adaptive manner. This includes psychological/behavioral strategies, mind-body approaches, lifestyle advice, pain education and pain coping.
  Arms: Supported-Self management (SSM)
Other: Spinal Manipulation Therapy (SMT) — SMT will address the biological and physical aspects of low back pain (e.g. spinal dysfunction) with the intention of restoring maximum movement and functional ability of the spine.
  Arms: Spinal Manipulation Therapy (SMT)
Combination Product: SMT + SSM — Combination Treatment
  Arms: SMT + SSM
Drug: Standard Medical Care (SMC) — Guideline based medical care informed by the American College of Physicians' guidelines on noninvasive treatment for low back pain.
  Arms: Standard Medical Care (SMC)

SUMMARY:
This is a study of adults with acute low back pain flare-up at risk of becoming chronic and disabling. The study tests how well spinal manipulation and guided selfcare work compared to standard medical care. The treatments last up to eight weeks and participants will be followed for one year.

DETAILED DESCRIPTION:
The long-term goal is to reduce overall low back pain (LBP) burden by evaluating, first-line, non-drug treatment strategies that address the biological, psychological and social aspects of acute LBP and prevent transition to chronic back pain. The study will also assess barriers and facilitators that impact future implementation of the non-drug treatments into clinical practice.

The US faces an unprecedented pain management crisis. LBP is the most common chronic pain condition in adults and one of the leading causes of disability worldwide. Guidelines have recommended non-drug treatments like spinal manipulation and behavioral and selfcare approaches for LBP for nearly a decade, yet uptake and adherence has been poor. Little is known about the role of these treatments in the secondary prevention of chronic LBP, especially for patients at risk of developing severe low back pain. Due to high societal costs, and side effects of commonly used drug treatments, including opioids, there is a critical need for research on how well non-drug treatments work for preventing serious chronic LBP.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Acute or sub-acute low back pain
* Average low back pain severity ≥3 on the 0-10 numerical rating scale over 7 days
* Medium or high risk for persistent disabling back pain according to the STarT Back screening tool
* Ability to read and write fluently in English

Exclusion Criteria:

* Non-mechanical causes of low back pain
* Contraindications to study treatments (e.g,. surgical fusion of lumbar spine)
* Active management of current episode of low back pain by another healthcare provider
* Serious co-morbid health condition that either requires medical attention or has a risk for general health decline over the next year
* Pregnancy, current or planned during study period and nursing mothers
* Inability or unwillingness to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gert Bronfort, PhD, DC, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - University of Minnesota, Minneapolis, Minnesota
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Bronfort G, Meier EN, Leininger B, Schneider M, Evans R, Greco C, Hanson L, McFarland C, Chou R, Connett J, Delitto A, George SZ, Glick RM, Keefe F, Licciardone J, Schulz C, Turk D, Heagerty PJ. Spinal Manipulation and Clinician-Supported Biopsychosocial Self-Management for Acute Back Pain: The PACBACK Randomized Clinical Trial. JAMA. 2025 Dec 29:e2521990. doi: 10.1001/jama.2025.21990. Online ahead of print. PMID 41460638
- [Derived] Bronfort G, Delitto A, Schneider M, Heagerty PJ, Chou R, Connett J, Evans R, George S, Glick RM, Greco C, Hanson L, Keefe F, Leininger B, Licciardone J, McFarland C, Meier E, Schulz C, Turk D. Effectiveness of spinal manipulation and biopsychosocial self-management compared to medical care for low back pain: a randomized trial study protocol. BMC Musculoskelet Disord. 2023 May 25;24(1):415. doi: 10.1186/s12891-023-06549-w. PMID 37231386
- [Derived] Bronfort G, Delitto A, Schneider M, Heagerty P, Chou R, Connett J, Evans R, George S, Glick R, Greco C, Hanson L, Keefe F, Leininger B, Licciardone J, McFarland C, Meier E, Schulz C, Turk D. Effectiveness of Spinal Manipulation and Biopsychosocial Self-Management compared to Medical Care for Low Back Pain: A Randomized Trial Study Protocol. Res Sq [Preprint]. 2023 May 3:rs.3.rs-2865633. doi: 10.21203/rs.3.rs-2865633/v1. PMID 37205428

RESULTS

PARTICIPANT FLOW:
Groups:
- Supported Self-Management (SSM): Supported Self-Management (SSM): Provides low back pain sufferers opportunities to develop the capacity and motivation to self-manage their pain in an adaptive manner. This includes psychological/behavioral strategies, mind-body approaches, lifestyle advice, pain education and pain coping.
- Spinal Manipulation Therapy (SMT): Spinal manipulation therapy (SMT): Addresses the biological and physical aspects of low back pain (e.g. spinal dysfunction) with the intention of restoring maximum movement and functional ability of the spine.
- Combined SSM/SMT: Supported self-management / spinal manipulation therapy (SSM/SMT): Combination treatment.
- Medical Care (MC): Medical care (MC): Guideline based medical care informed by the American College of Physicians' guidelines on noninvasive treatment for low back pain.
Period: Treatment Adherence Assessment
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Started | 305 | 201 | 193 | 301
Adherent to Treatment | 271 | 168 | 156 | 290
Non-adherent, Due to COVID (Adherence was defined as attending at least 2 visits (4 for SSM), not missing more than 25% of scheduled visits, and not dropping out of active care. Participants who failed to meet one or more of these criteria due to COVID or COVID protocols are listed in this row.) | 4 | 19 | 18 | 2
Non-adherent, Not Due to COVID (Adherence was defined as attending at least 2 visits (4 for SSM), not missing more than 25% of scheduled visits, and not dropping out of active care. Participants who failed to meet one or more of these criteria for reasons other than COVID or COVID protocols are listed in this row.) | 30 | 14 | 19 | 9
Completed | 305 | 201 | 193 | 301
Not Completed | 0 | 0 | 0 | 0
Period: 2-month Follow-up
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Started | 305 | 201 | 193 | 301
Completed Follow-up | 290 | 195 | 182 | 292
Missed Follow-up (Timed Out) | 2 | 1 | 3 | 3
Completed | 292 | 196 | 185 | 295
Not Completed | 13 | 5 | 8 | 6
Not completed — Withdrawal by Subject | 5 | 4 | 6 | 4
Not completed — Lost to Follow-up | 8 | 1 | 2 | 2
Period: 6-Month Follow-up
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Started | 292 | 196 | 185 | 295
Completed Follow-up | 282 | 188 | 180 | 284
Missed Follow-up (Timed Out) | 5 | 5 | 3 | 8
Completed | 287 | 193 | 183 | 292
Not Completed | 5 | 3 | 2 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 2
Not completed — Lost to Follow-up | 3 | 3 | 1 | 1
Period: 12-Month Follow-up
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Started | 287 | 193 | 183 | 292
Completed Follow-up | 280 | 187 | 178 | 283
Missed Follow-up (Timed Out) | 3 | 3 | 1 | 4
Completed | 283 | 190 | 179 | 287
Not Completed | 4 | 3 | 4 | 5
Not completed — Lost to Follow-up | 4 | 3 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC) | Total
Number analyzed (Participants) | 305 | 201 | 193 | 301 | 1000
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at randomization
  Years | 47 (15) | 48 (16) | 47 (17) | 47 (16) | 47 (16)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 175 | 104 | 117 | 181 | 577
  Gender: Male | 124 | 95 | 74 | 117 | 410
  Gender: Other | 5 | 2 | 2 | 3 | 12
  Gender: Unknown/not reported | 1 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 12 | 18 | 46
  Not Hispanic or Latino | 297 | 191 | 178 | 283 | 949
  Unknown or Not Reported | 1 | 1 | 3 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 2
  Asian | 17 | 11 | 13 | 18 | 59
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 25 | 7 | 16 | 18 | 66
  White | 258 | 172 | 154 | 251 | 835
  More than one race | 3 | 7 | 8 | 10 | 28
  Unknown or Not Reported | 1 | 4 | 2 | 3 | 10
Site [Count of Participants; unit: Participants]
  Minneapolis | 185 | 110 | 105 | 182 | 582
  Pittsburgh | 120 | 91 | 88 | 119 | 418
STarT Back Risk Category [Count of Participants; unit: Participants] — Risk stratification from the STarT Back Screening Tool
  Participants
    Medium | 212 | 150 | 135 | 202 | 699
    High | 93 | 51 | 58 | 99 | 301
Recruitment Time Period [Count of Participants; unit: Participants] — Due to COVID, the study was temporarily modified such that participants were randomized into only two arms that could be administered remotely (SSM and MC). We introduced a categorical time period measure to delineate three groups: participants randomized prior to the 2-arm period (pre-COVID), participants randomized during the 2-arm period (COVID), and participants randomized when the 4-arm period was resumed (post-COVID).
  Participants
    Pre-COVID | 46 | 47 | 48 | 45 | 186
    COVID | 106 | 0 | 0 | 105 | 211
    Post-COVID | 153 | 154 | 145 | 151 | 603
Pain intensity [Mean (Standard Deviation); unit: score on a scale] — Measured using the 0-10 numerical rating scale (0=no LBP, 10=the worst LBP possible).
  score on a scale | 5.5 (1.6) | 5.4 (1.5) | 5.4 (1.6) | 5.4 (1.6) | 5.4 (1.6)
Disability [Mean (Standard Deviation); unit: score on a scale] — Measured using the Roland-Morris Disability Questionnaire (RMDQ), a 24-item questionnaire that measures the degree to which a low back problem restricts daily activities. Score ranges from 0 to 24 with higher values indicating more disability.
  score on a scale | 11.6 (4.9) | 10.9 (4.6) | 10.8 (4.8) | 11.4 (4.5) | 11.2 (4.7)
Low Back Pain Impact Score [Mean (Standard Deviation); unit: score on a scale] — The LBP Impact Scale includes measures of pain intensity, pain interference, and physical function from the PROMIS-29 Profile v2.0. The scale ranges from 8 (least impact) to 50 (greatest impact).
  score on a scale | 25.9 (6.7) | 24.6 (6.6) | 25.2 (6.5) | 26.1 (6.7) | 25.6 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: Measured using the 0-10 numerical rating scale (0=no LBP, 10=the worst LBP possible). Missing weekly outcomes were multiply imputed. Means were estimated using marginal standardization with adjustment for site, time period, risk of chronicity, and baseline pain intensity.
Time Frame: Average over weeks 1-52
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 305 | 201 | 193 | 301
score on a scale | 2.8 (0.1) | 3.0 (0.1) | 2.8 (0.1) | 3.0 (0.1)
Statistical Analysis 1: Comparison: Supported Self-Management (SSM) vs Spinal Manipulation Therapy (SMT) vs Combined SSM/SMT vs Medical Care (MC); The null hypothesis here is that the means are equal across the 4 treatment groups. A significant p value indicates rejection of the null; Test type: Other — Omnibus test for equality of means across the 4 treatment groups; p = 0.16, ANOVA — Threshold for significance: 0.025 (0.05/2); Adjusted for site, time period (pre-COVID, COVID, post-COVID), risk for chronicity (medium vs. high), and baseline pain intensity
Statistical Analysis 2: Comparison: Supported Self-Management (SSM) vs Medical Care (MC); Adjusted for site, time period, risk of chronicity, and baseline pain intensity; Test type: Other — Estimation; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.5 to 0.0] — SSM - MC
Statistical Analysis 3: Comparison: Spinal Manipulation Therapy (SMT) vs Medical Care (MC); Adjusted for site, time period, risk of chronicity, and baseline pain intensity; Test type: Other — Estimation; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.3 to 0.3] — SMT - MC
Statistical Analysis 4: Comparison: Combined SSM/SMT vs Medical Care (MC); Adjusted for site, time period, risk of chronicity, and baseline pain intensity; Test type: Other — Estimation; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.4 to 0.1] — SSM/SMT - MC

2. Primary Outcome: Disability
Description: Measured using the Roland-Morris Disability Questionnaire (RMDQ), a 24-item questionnaire that measures the degree to which a low back problem restricts daily activities. Score ranges from 0 to 24 with higher values indicating more disability. Missing monthly outcomes were multiply imputed. Means were estimated using marginal standardization with adjustment for site, time period, risk of chronicity, and baseline RMDQ.
Time Frame: Average over months 1-12
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 305 | 201 | 193 | 301
score on a scale | 4.7 (0.2) | 5.5 (0.3) | 4.8 (0.3) | 5.9 (0.2)
Statistical Analysis 1: Comparison: Supported Self-Management (SSM) vs Spinal Manipulation Therapy (SMT) vs Combined SSM/SMT vs Medical Care (MC); [analysis description as in outcome 1, analysis 1]; Test type: Other — Omnibus test for equality of means across the 4 treatment groups; p = 0.001, ANOVA — Threshold for significance: 0.025 (0.05/2); Adjusted for site, time period (pre-COVID, COVID, post-COVID), risk for chronicity (medium vs. high), and baseline disability
Statistical Analysis 2: Comparison: Supported Self-Management (SSM) vs Medical Care (MC); Adjusted for site, time period, risk of chronicity, and baseline RMDQ; Test type: Other — Estimation; Mean Difference (Net) = -1.2, 95% CI 2-sided [-1.9 to -0.5] — SSM - MC
Statistical Analysis 3: Comparison: Spinal Manipulation Therapy (SMT) vs Medical Care (MC); Adjusted for site, time period, risk of chronicity, and baseline RMDQ; Test type: Other — Estimation; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.2 to 0.4] — SMT - MC
Statistical Analysis 4: Comparison: Combined SSM/SMT vs Medical Care (MC); Adjusted for site, time period, risk of chronicity, and baseline RMDQ; Test type: Other — Estimation; Mean Difference (Net) = -1.1, 95% CI 2-sided [-1.9 to -0.3] — SSM/SMT - MC

3. Primary Outcome: Low Back Pain (LBP) That is Impactful
Description: Measured by the LBP impact scale, which includes measures of pain intensity, pain interference, and physical function from the PROMIS-29 Profile v2.0. The scale ranges from 8 (least impact) to 50 (greatest impact). Missing monthly outcomes were multiply imputed. Means were estimated using marginal standardization with adjustment for site, time period, risk of chronicity, and baseline LBP impact score.
Time Frame: Average over months 10 -12
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 305 | 201 | 193 | 301
score on a scale | 15.3 (0.4) | 16.7 (0.5) | 15.7 (0.5) | 17.0 (0.4)
Statistical Analysis 1: Comparison: Supported Self-Management (SSM) vs Spinal Manipulation Therapy (SMT) vs Combined SSM/SMT vs Medical Care (MC); [analysis description as in outcome 1, analysis 1]; Test type: Other — Omnibus test for equality of means across the 4 treatment groups; p = 0.006, ANOVA — Threshold for significance: 0.05; Adjusted for site, time period (pre-COVID, COVID, post-COVID), risk for chronicity (medium vs. high), and baseline LBP impact score
Statistical Analysis 2: Comparison: Supported Self-Management (SSM) vs Medical Care (MC); Adjusted for site, time period, risk of chronicity, and baseline LBP impact score; Test type: Other — Estimation; Mean Difference (Net) = -1.7, 95% CI 2-sided [-2.7 to -0.6] — SSM - MC
Statistical Analysis 3: Comparison: Spinal Manipulation Therapy (SMT) vs Medical Care (MC); Adjusted for site, time period, risk of chronicity, and baseline LBP impact score; Test type: Other — Estimation; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.5 to 1.0] — SMT - MC
Statistical Analysis 4: Comparison: Combined SSM/SMT vs Medical Care (MC); Adjusted for site, time period, risk of chronicity, and baseline LBP impact score; Test type: Other — Estimation; Mean Difference (Net) = -1.3, 95% CI 2-sided [-2.5 to -0.0] — SSM/SMT - MC

4. Secondary Outcome: Recovery From Acute/Sub-acute Low Back Pain
Description: Measured by the proportion of patients with scores of 0 on the 0-10 pain numeric rating scale (NRS) and a score of less than or equal to 2 on the Roland-Morris Disability Questionnaire (RMDQ), a 24-item questionnaire that measures the degree to which a low back problem restricts daily activities.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 282 | 186 | 177 | 284
Participants | 56 | 29 | 33 | 38

5. Secondary Outcome: Low Back Pain Frequency - Percent of Days Over 12 Months
Description: Participants report the number of days that low back pain has been a problem in the past 7 days for 52 weeks. This measure is the percent of days that low back pain has been a problem. Mean and confidence intervals are estimated using marginal standardization and bootstrapping. Adjustment for site, time period, and risk for chronicity.
Time Frame: Weeks 1-52
Population: Only participants with at least 35 weeks of follow-up between weeks 1 and 52 are included in the analysis.
Measure: Mean (95% Confidence Interval); unit: Percent of days
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 273 | 185 | 173 | 281
Percent of days | 39 [36 to 43] | 44 [40 to 48] | 38 [34 to 42] | 46 [42 to 49]
Statistical Analysis 1: Comparison: Supported Self-Management (SSM) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percent difference); Risk Difference (RD) = -6, 95% CI 2-sided [-11 to -1] — SSM - MC
Statistical Analysis 2: Comparison: Spinal Manipulation Therapy (SMT) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -1, 95% CI 2-sided [-7 to 5] — SMT - MC
Statistical Analysis 3: Comparison: Combined SSM/SMT vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -8, 95% CI 2-sided [-13 to 2] — SSM/SMT - MC

6. Secondary Outcome: Number of Participants Who Received Care For Low Back Pain
Description: Includes provider visits, emergency department visits, diagnostic imaging scans, hospitalizations, injections and surgical procedures. This is a binary indicator of any care from providers outside the study for low back pain.
Time Frame: Months 1-12
Population: Only participants with at least 8 months of follow-up between months 1 and 12 on this outcome are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 277 | 187 | 178 | 283
Participants | 82 | 67 | 53 | 128
Statistical Analysis 1: Comparison: Supported Self-Management (SSM) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -15, 95% CI 2-sided [-23 to -7] — SSM - MC
Statistical Analysis 2: Comparison: Spinal Manipulation Therapy (SMT) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -11, 95% CI 2-sided [-20 to 2] — SMT - MC
Statistical Analysis 3: Comparison: Combined SSM/SMT vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -18, 95% CI 2-sided [-27 to -9] — SSM/SMT - MC

7. Secondary Outcome: Medication Use - Percent of Months 4-12
Description: Over the counter and prescription medication use for low back pain. Since the MC arm intervention includes medications, only months 4-12 (i.e. after the intervention) are considered for this outcome. The measure is the percent of months 4-12 in which medication was used for low back pain. Mean and confidence intervals are estimated using marginal standardization and bootstrapping. Adjustment for site, time period, and risk for chronicity.
Time Frame: Months 4-12
Population: Only participants with at least 6 months of follow-up between months 4 and 12 are included in the analysis.
Measure: Mean (95% Confidence Interval); unit: Percent of months 4-12
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 277 | 188 | 179 | 283
Percent of months 4-12 | 37 [33 to 42] | 40 [34 to 46] | 37 [31 to 43] | 54 [50 to 58]
Statistical Analysis 1: Comparison: Supported Self-Management (SSM) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -16, 95% CI 2-sided [-23 to -10] — SSM - MC
Statistical Analysis 2: Comparison: Spinal Manipulation Therapy (SMT) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -14, 95% CI 2-sided [-22 to -7] — SMT - MC
Statistical Analysis 3: Comparison: Combined SSM/SMT vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -17, 95% CI 2-sided [-24 to -9] — SSM/SMT - MC

8. Secondary Outcome: Bothered by Low Back Pain at Work - Percent of Months
Description: Participants indicated in monthly follow-ups if they were bothered by low back pain over the last month. This measure is the percent of months that participants were bothered by low back pain at work. Mean and confidence intervals are estimated using marginal standardization and bootstrapping. Adjustment for site, time period, and risk for chronicity.
Time Frame: Months 1-12
Population: Only participants with at least 8 months of follow-up between months 1 and 12 are included in the analysis.
Measure: Mean (95% Confidence Interval); unit: Percent of months
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 279 | 189 | 179 | 285
Percent of months | 43 [39 to 47] | 45 [40 to 51] | 43 [38 to 48] | 51 [47 to 55]
Statistical Analysis 1: Comparison: Supported Self-Management (SSM) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -8, 95% CI 2-sided [-13 to -3] — SSM - MC
Statistical Analysis 2: Comparison: Spinal Manipulation Therapy (SMT) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -5, 95% CI 2-sided [-12 to 1] — SMT - MC
Statistical Analysis 3: Comparison: Combined SSM/SMT vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -8, 95% CI 2-sided [-15 to -1] — SSM/SMT - MC

9. Secondary Outcome: Global Improvement
Description: Measured using a 9-point scale: 0 (vastly worse) to 8 (completely recovered )
Time Frame: 2 months
Population: The Participant Flow tables show counts of completed follow-up defined by completion of the Roland-Morris Disability Questionnaire (RMDQ). There are some participants who completed the RMDQ but not this measure and vice versa. Thus the analysis counts for each time point here may differ somewhat from the Participant Flow tables.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 290 | 193 | 183 | 291
score on a scale | 6.2 (1.2) | 6.3 (1.0) | 6.4 (1.1) | 5.7 (1.5)

10. Secondary Outcome: Global Improvement
Description: Measured using a 9-point scale: 0 (vastly worse) to 8 (completely recovered )
Time Frame: 6 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 281 | 187 | 178 | 281
score on a scale | 6.1 (1.4) | 6.0 (1.3) | 6.3 (1.4) | 5.5 (1.7)

11. Secondary Outcome: Global Improvement
Description: Measured using a 9-point scale: 0 (vastly worse) to 8 (completely recovered )
Time Frame: 12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 279 | 187 | 177 | 280
score on a scale | 6.2 (1.3) | 5.8 (1.6) | 6.3 (1.4) | 5.5 (1.6)

12. Secondary Outcome: Patient Satisfaction With Treatment
Description: Measured using a 7-point Likert scale: 0 (completely dissatisfied) to 6 (completely satisfied)
Time Frame: 2 months
Population: The counts above are for participants that completed the satisfaction question at the 2-month time point. The Participant Flow tables show counts of completed follow-up defined by completion of the Roland-Morris Disability Questionnaire (RMDQ). There are some participants who completed the RMDQ but not this measure and vice versa. Thus the analysis counts for each time point here may differ somewhat from the Participant Flow tables.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 289 | 193 | 183 | 291
score on a scale | 4.9 (1.0) | 5.0 (0.9) | 5.2 (0.9) | 4.2 (1.3)

13. Secondary Outcome: Patient Satisfaction With Treatment
Description: Measured using a 7-point Likert scale: 0 (completely dissatisfied) to 6 (completely satisfied)
Time Frame: 6 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 281 | 188 | 177 | 281
score on a scale | 4.8 (1.0) | 4.8 (1.1) | 5.1 (0.9) | 4.1 (1.4)

14. Secondary Outcome: Patient Satisfaction With Treatment
Description: Measured using a 7-point Likert scale: 0 (completely dissatisfied) to 6 (completely satisfied)
Time Frame: 12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 279 | 183 | 177 | 281
score on a scale | 4.7 (1.1) | 4.6 (1.1) | 5.1 (1.0) | 4.0 (1.4)

15. Secondary Outcome: Chronic Low Back Pain (LBP)
Description: Measured by the proportion of patients in each group meeting the definition by the NIH Task Force on Research Standards for Chronic LBP (i.e., ongoing LBP on ≥50% of days over past 6 months).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 280 | 186 | 178 | 279
Participants | 119 | 81 | 78 | 154
Statistical Analysis 1: Comparison: Supported Self-Management (SSM) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -12, 95% CI 2-sided [-21 to -4] — SSM - MC
Statistical Analysis 2: Comparison: Spinal Manipulation Therapy (SMT) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -12, 95% CI 2-sided [-22 to -3] — SMT - MC
Statistical Analysis 3: Comparison: Combined SSM/SMT vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -12, 95% CI 2-sided [-22 to -3] — SSM/SMT - MC

16. Secondary Outcome: Chronic Low Back Pain (LBP)
Description: as for outcome 15
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 277 | 185 | 177 | 282
Participants | 93 | 93 | 68 | 151
Statistical Analysis 1: Comparison: Supported Self-Management (SSM) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -20, 95% CI 2-sided [-28 to -12] — SSM - MC
Statistical Analysis 2: Comparison: Spinal Manipulation Therapy (SMT) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -4, 95% CI 2-sided [-13 to 6] — SMT - MC
Statistical Analysis 3: Comparison: Combined SSM/SMT vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -16, 95% CI 2-sided [-26 to -7] — SSM/SMT - MC

17. Secondary Outcome: Number of Participants Who Reported Chronic Interference With Daily Activities
Description: Assessed using "how often has low back pain interfered with your ability to do regular activities over the past 6 months?" on a 3-item scale (less than half the days in the past 6 months, at least half the days in the past 6 months, every day or nearly every day in the past 6 months). Here we dichotomize to "at least half the days in the past 6 months" or more.
Time Frame: 6 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 279 | 185 | 179 | 282
Participants | 57 | 41 | 38 | 80
Statistical Analysis 1: Comparison: Supported Self-Management (SSM) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -8, 95% CI 2-sided [-15 to -1] — SSM - MC
Statistical Analysis 2: Comparison: Spinal Manipulation Therapy (SMT) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -7, 95% CI 2-sided [-22 to -3] — SMT - MC
Statistical Analysis 3: Comparison: Combined SSM/SMT vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -12, 95% CI 2-sided [-22 to -3] — SSM/SMT - MC

18. Secondary Outcome: Number of Participants Who Reported Chronic Interference With Daily Activities
Description: as for outcome 17
Time Frame: 12 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 278 | 187 | 177 | 281
Participants | 41 | 36 | 36 | 76
Statistical Analysis 1: Comparison: Supported Self-Management (SSM) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -12, 95% CI 2-sided [-19 to -5] — SSM - MC
Statistical Analysis 2: Comparison: Spinal Manipulation Therapy (SMT) vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -8, 95% CI 2-sided [-16 to -1] — SMT - MC
Statistical Analysis 3: Comparison: Combined SSM/SMT vs Medical Care (MC); Adjusted for site, time period, and risk of chronicity; Test type: Other — Estimation (percentage difference); Risk Difference (RD) = -8, 95% CI 2-sided [-16 to 1] — SSM/SMT - MC

19. Secondary Outcome: Timed Up and Go Test
Description: Measured by a blinded examiner, in seconds, the time taken by a person to stand up, walk a distance of 10 feet, turn, walk back to the chair and sit down again.
Time Frame: 2 months
Population: Unlike outcomes collected via surveys, this outcome required an in-person meeting or teleconference. It was frequently difficult to schedule within the outcome window and thus has lower follow-up than survey outcomes.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 243 | 167 | 152 | 242
seconds | 9.5 (2.0) | 9.5 (2.3) | 9.5 (3.0) | 10.0 (2.2)

20. Secondary Outcome: Sit-to-stand
Description: Measured by a blinded examiner, in seconds, the amount of time a person requires to stand up and sit down from a chair 5 times without using their arms
Time Frame: 2 months
Population: Unlike outcomes collected via surveys, this outcome required an in-person meeting or teleconference. It was frequently difficult to schedule within the outcome window and thus has lower follow-up than survey outcomes. Measure was not collected in the UG3 phase of the study (November 2018 through April 2019).
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 223 | 146 | 132 | 223
seconds | 10.5 (2.8) | 11.4 (3.3) | 10.9 (2.9) | 10.9 (3.4)

21. Secondary Outcome: The Sock Test
Description: Measured by a blinded examiner on a scale from 0-3, with 0 being can easily grab the toes with the fingertips of both hands and 3 being can hardly, if at all, reach as far as to the malleoli. Each leg is scored separately with the greater leg score serving as the overall score.
Time Frame: 2 months
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 237 | 166 | 152 | 244
Participants
  0: Patient can easily reach and grab toes with fingertips. | 112 | 65 | 53 | 114
  1: Patient can reach toes with effort. | 28 | 15 | 17 | 30
  2: Patient can reach beyond the malleoli but cannot reach toes. | 20 | 23 | 28 | 25
  3: Patient has difficulty reaching even the malleoli. | 77 | 63 | 54 | 75

22. Secondary Outcome: Visual Trajectory for Pain
Description: Assessed using 8 different diagrams describing back pain change over the last 12 months
Time Frame: 12 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 277 | 186 | 178 | 282
Participants
  (a) A single episode with no other major episode of back pain | 18 | 6 | 13 | 15
  (b) A few episodes of back pain, with mostly pain-free periods in between | 103 | 53 | 51 | 65
  (c) Some back pain most of the time, and a few episodes of severe pain | 72 | 58 | 56 | 99
  (d) Pain that goes up and down all the time, with episodes of severe back pain | 26 | 25 | 16 | 51
  (e) Severe back pain all or nearly all of the time | 2 | 2 | 0 | 6
  (f) Back pain that has got gradually worse | 2 | 2 | 3 | 3
  (g) Back pain that has improved gradually | 38 | 28 | 28 | 33
  (h) No back pain, or only the odd day with mild pain | 16 | 12 | 11 | 10

23. Secondary Outcome: Quebec Task Force
Description: Measured by a blinded examiner who will classify the participant's spinal disorder as 0) no pain; 1) pain without radiation; 2) pain with radiation to the proximal extremity; 3) pain with radiation to the distal extremity; 4) pain with radiation to the extremity and neurologic signs.
Time Frame: 2 months
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 248 | 167 | 155 | 253
Participants
  0: No pain | 70 | 38 | 32 | 59
  1: Pain without radiation | 150 | 106 | 100 | 163
  2: Pain with radiation to extremity, proximally | 19 | 10 | 11 | 13
  3: Pain with radiation to extremity, distally | 8 | 13 | 10 | 13
  4: Pain with radiation to lower limb with neurologic signs | 1 | 0 | 2 | 5

24. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Depression
Description: The PROMIS depression scale consists of 4 questions related to depression over the past 7 days. The raw score is converted to the T-Score that is reported here. The range of possible scores is 41.0 - 79.3. Higher scores indicate greater depression. A score of 50 represents the average score in a general US reference population and 10 is the standard deviation.
Time Frame: Baseline and 2, 6, and 12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 305 | 201 | 193 | 301
T-Score
  Baseline | 50.6 (7.2) | 50.2 (7.4) | 50.8 (7.3) | 50.8 (8.3)
  2-month: number analyzed (Participants) | 290 | 195 | 183 | 292
  2-month | 49.6 (7.6) | 49.0 (7.9) | 49.7 (8.2) | 50.4 (8.0)
  6-month: number analyzed (Participants) | 282 | 188 | 180 | 283
  6-month | 48.2 (8.1) | 48.2 (7.8) | 48.6 (8.4) | 49.6 (8.5)
  12-month: number analyzed (Participants) | 280 | 187 | 178 | 283
  12-month | 48.2 (8.0) | 47.8 (8.2) | 48.2 (8.2) | 49.0 (8.9)

25. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function
Description: The PROMIS physical function scale consists of 4 questions about ability to perform tasks of daily living. The raw score is converted to the T-Score that is reported here. The range of possible scores is 22.6 - 57.0. Higher scores indicate greater physical function. A score of 50 represents the average score in a general US reference population and 10 is the standard deviation.
Time Frame: Baseline and 2, 6, and 12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 305 | 201 | 193 | 301
T-Score
  Baseline | 40.7 (4.6) | 21.7 (5.7) | 41.3 (5.5) | 40.5 (4.9)
  2-month: number analyzed (Participants) | 290 | 195 | 183 | 292
  2-month | 46.0 (6.8) | 46.8 (7.3) | 46.4 (7.0) | 44.8 (6.9)
  6-month: number analyzed (Participants) | 282 | 188 | 180 | 284
  6-month | 48.0 (7.5) | 47.3 (7.4) | 47.5 (8.1) | 46.3 (7.6)
  12-month: number analyzed (Participants) | 280 | 187 | 177 | 284
  12-month | 48.5 (7.5) | 47.7 (7.7) | 48.6 (7.7) | 46.6 (7.4)

26. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Anxiety
Description: The PROMIS anxiety scale consists of 4 questions related to anxiety over the past 7 days. The raw score is converted to the T-Score that is reported here. The range of possible scores is 40.3 - 81.4. Higher scores indicate greater anxiety. A score of 50 represents the average score in a general US reference population and 10 is the standard deviation.
Time Frame: Baseline and 2, 6, and 12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 305 | 201 | 193 | 301
T-Score
  Baseline | 53.5 (8.2) | 53.6 (7.9) | 54.2 (7.6) | 53.8 (8.3)
  2-month: number analyzed (Participants) | 290 | 195 | 183 | 292
  2-month | 51.7 (8.0) | 51.2 (8.2) | 52.6 (8.3) | 52.6 (8.5)
  6-month: number analyzed (Participants) | 282 | 188 | 180 | 283
  6-month | 49.4 (8.9) | 49.2 (9.2) | 50.6 (9.7) | 50.3 (9.5)
  12-month: number analyzed (Participants) | 280 | 187 | 177 | 283
  12-month | 48.9 (9.1) | 48.7 (8.9) | 49.1 (9.5) | 50.1 (9.8)

27. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Fatigue
Description: The PROMIS fatigue scale consists of 4 questions related to fatigue over the past 7 days. The raw score is converted to the T-Score that is reported here. The range of possible scores is 33.7 - 75.8. Higher scores indicate greater fatigue. A score of 50 represents the average score in a general US reference population and 10 is the standard deviation.
Time Frame: Baseline and 2, 6, and 12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 305 | 201 | 193 | 301
T-Score
  Baseline | 55.2 (8.1) | 54.3 (8.1) | 54.8 (8.0) | 55.2 (8.5)
  2-month: number analyzed (Participants) | 290 | 195 | 183 | 292
  2-month | 52.4 (8.5) | 51.2 (8.0) | 51.8 (8.4) | 53.8 (9.2)
  6-month: number analyzed (Participants) | 282 | 188 | 180 | 283
  6-month | 51.3 (9.7) | 50.8 (9.7) | 50.4 (10.1) | 52.2 (10.5)
  12-month: number analyzed (Participants) | 280 | 187 | 178 | 283
  12-month | 50.8 (10.1) | 50.6 (10.1) | 50.0 (10.2) | 52.3 (10.1)

28. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance
Description: The PROMIS sleep disturbance scale consists of 4 questions related to sleep disturbance over the past 7 days. The raw score is converted to the T-Score that is reported here. The range of possible scores is 32.0 - 73.3. Higher scores indicate greater sleep disturbance. A score of 50 represents the average score in a general US reference population and 10 is the standard deviation.
Time Frame: Baseline and 2, 6, and 12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 305 | 201 | 193 | 301
T-Score
  Baseline | 52.0 (3.0) | 51.8 (3.4) | 52.0 (3.5) | 52.1 (3.1)
  2-month: number analyzed (Participants) | 290 | 195 | 183 | 292
  2-month | 52.6 (3.1) | 52.2 (2.9) | 52.1 (3.8) | 52.2 (3.0)
  6-month: number analyzed (Participants) | 282 | 188 | 180 | 283
  6-month | 52.2 (3.6) | 51.8 (3.7) | 52.1 (3.5) | 51.9 (3.4)
  12-month: number analyzed (Participants) | 280 | 187 | 178 | 283
  12-month | 52.2 (3.0) | 52.1 (3.3) | 51.7 (3.6) | 51.7 (3.7)

29. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Participation
Description: The PROMIS participation scale consists of 4 questions related to participation in social activities. The raw score is converted to the T-Score that is reported here. The range of possible scores is 27.5 - 64.2. Higher scores indicate greater ability to participate in social activities. A score of 50 represents the average score in a general US reference population and 10 is the standard deviation.
Time Frame: Baseline and 2, 6, and 12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 305 | 201 | 193 | 301
T-Score
  Baseline | 46.8 (6.1) | 47.7 (6.7) | 47.7 (7.2) | 46.6 (6.0)
  2-month: number analyzed (Participants) | 290 | 195 | 183 | 292
  2-month | 53.2 (7.6) | 53.5 (7.4) | 52.9 (7.7) | 52.1 (8.0)
  6-month: number analyzed (Participants) | 282 | 188 | 180 | 283
  6-month | 54.8 (7.9) | 54.5 (8.5) | 55.0 (8.7) | 53.5 (8.4)
  12-month: number analyzed (Participants) | 280 | 187 | 178 | 283
  12-month | 55.2 (8.0) | 54.7 (8.4) | 55.8 (8.4) | 54.1 (8.5)

30. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference
Description: The PROMIS participation scale consists of 4 questions related to pain interference in the last 7 days. The raw score is converted to the T-Score that is reported here. The range of possible scores is 41.6 - 75.6. Higher scores indicate greater pain interference. A score of 50 represents the average score in a general US reference population and 10 is the standard deviation.
Time Frame: Baseline and 2, 6, and 12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 305 | 201 | 193 | 301
T-Score
  Baseline | 60.3 (5.0) | 59.2 (5.4) | 59.9 (5.3) | 60.3 (5.2)
  2-month: number analyzed (Participants) | 290 | 195 | 183 | 292
  2-month | 52.9 (7.0) | 52.0 (7.3) | 52.4 (7.3) | 53.9 (7.8)
  6-month: number analyzed (Participants) | 282 | 188 | 180 | 283
  6-month | 51.4 (7.9) | 51.5 (7.6) | 51.2 (8.0) | 52.7 (8.3)
  12-month: number analyzed (Participants) | 280 | 187 | 178 | 283
  12-month | 50.3 (8.4) | 51.0 (7.9) | 50.6 (7.9) | 52.4 (8.0)

31. Secondary Outcome: STarT Back Risk Classification
Description: The STarT Back Screening Tool is a 9-item questionnaire used to identify prognostic risk factors in patients with low back pain. It assesses physical and psychosocial factors, including referred pain, disability, fear-avoidance, anxiety, and depression. Scores are totaled (0-9) and a psychosocial subscale score (items 5-9, range 0-5) is calculated. Patients are classified as: low risk (total ≤3), medium risk (total ≥4 and psychosocial subscale ≤3), or high risk (total ≥4 and psychosocial subscale ≥4).
Time Frame: 2 months
Population: The Participant Flow tables show counts of completed follow-up defined by completion of the Roland-Morris Disability Questionnaire (RMDQ). There are some participants who completed the RMDQ but not this measure and vice versa. Thus the analysis counts may differ somewhat from the Participant Flow tables.
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 289 | 194 | 182 | 291
Participants
  Low risk | 238 | 164 | 160 | 226
  Medium risk | 45 | 28 | 19 | 46
  High risk | 6 | 2 | 3 | 19

32. Secondary Outcome: STarT Back Risk Classification
Description: as for outcome 31
Time Frame: 6 months
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 281 | 186 | 179 | 283
Participants
  Low risk | 253 | 156 | 147 | 214
  Medium risk | 23 | 24 | 27 | 55
  High risk | 5 | 6 | 5 | 14

33. Secondary Outcome: STarT Back Risk Classification
Description: as for outcome 31
Time Frame: 12 months
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
Number analyzed (Participants) | 280 | 186 | 178 | 279
Participants
  Low risk | 243 | 158 | 157 | 226
  Medium risk | 34 | 23 | 18 | 39
  High risk | 3 | 5 | 3 | 14

34. Other Pre Specified Outcome: Self-efficacy
Description: Using a 10-100 numerical rating scale (10=very uncertain, 100 = very certain), self-efficacy is measured with the 22-item Chronic Pain Self-Efficacy Scale adapted for acute/sub-acute pain. This is a psychosocial mediating measure.
Time Frame: Baseline, 2, 6, 12 months
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Catastrophizing
Description: Measured using the 13-item Pain Catastrophizing Scale; it uses a 5-item point scale (0=not at all, 4 all the time). This is a psychosocial mediating measure.
Time Frame: Baseline, 2, 6, 12 months
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Kinesiophobia
Description: Measured using the 11-item Tampa Scale for Kinesiophobia demonstrated to have internal consistency, responsiveness and validity similar to the original 17-item instrument. A four-item scale is used (strongly disagree to strongly agree). This is a psychosocial mediating measure.
Time Frame: Baseline, 2, 6, 12 months
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Coping
Description: Measured using an adapted version of the 28-item Brief Coping Orientation to Problems Experienced (COPE) instrument on a 4 point scale (I haven't been doing this at all to I've been doing this a lot). This is a psychosocial mediating measure.
Time Frame: Baseline, 2, 6, 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year from randomization
Description: Participants were queried about adverse events during treatment visits and in all monthly surveys. Participants who did not have any treatment visits are excluded from the adverse events tabulations. Thus denominators differ from the overall study population.
Arm/Group | Supported Self-Management (SSM) | Spinal Manipulation Therapy (SMT) | Combined SSM/SMT | Medical Care (MC)
All-Cause Mortality (participants affected / at risk) | 0/298 | 0/198 | 0/190 | 0/296
Serious Adverse Events (participants affected / at risk) | 27/298 | 13/198 | 22/190 | 22/296
Other Adverse Events (participants affected / at risk) | 93/298 | 63/198 | 63/190 | 82/296
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supported Self-Management (SSM) (N=298) | Spinal Manipulation Therapy (SMT) (N=198) | Combined SSM/SMT (N=190) | Medical Care (MC) (N=296)
Lumbar back-related procedure (Surgical and medical procedures) | 2 (2) | 0 (0) | 2 (2) | 3 (3)
Other surgical/medical procedure (Surgical and medical procedures) | 6 (6) | 7 (8) | 6 (8) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fall or accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
COVID (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Non-COVID infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Inpatient mental health visit (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac problems (Cardiac disorders) | 2 (2) | 1 (1) | 3 (3) | 4 (4)
Diabetes complications (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal issues (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (3) | 1 (1)
Respiratory issue (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancers (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nervous system problem (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Severe vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fluid retention in abdomen and lungs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice from gallstones (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylaxis from known allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inpatient diagnostic visit (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition due to anorexia nervosa (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thumb pain/weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine blood clot (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood clot in lung (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hospitalization without additional information (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supported Self-Management (SSM) (N=298) | Spinal Manipulation Therapy (SMT) (N=198) | Combined SSM/SMT (N=190) | Medical Care (MC) (N=296)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (25) | 15 (17) | 19 (23) | 42 (52)
COVID (Infections and infestations) | 38 (40) | 35 (37) | 21 (22) | 25 (26)
Non-COVID infection (Infections and infestations) | 29 (35) | 14 (16) | 21 (23) | 13 (15)
Gastrointestinal issues (Gastrointestinal disorders) | 20 (23) | 12 (12) | 18 (21) | 16 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT03581123/Prot_SAP_000.pdf